CLINICAL TRIAL: NCT06494839
Title: Outcomes of Bipolar Electrocautery Tonsillectomy Versus Cold Steel Dissection Pediatric Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TonsillectomyLHR
Record Dates: First submitted 2024-06-26; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bipolar electrocautery tonsillectomy group (Experimental)
  Interventions: Procedure: Bipolar electrocautery tonsillectomy technique
- Cold steel dissection group (Experimental)
  Interventions: Procedure: Cold steel dissection technique

INTERVENTIONS:
Procedure: Bipolar electrocautery tonsillectomy technique — The BED tonsillectomy procedures were done under general anesthesia, and the patient's position was the same as in the other method. The bipolar machine was adjusted to 30 watts, and a mucosal incision was cauterized with a single straight or stepped bipolar forceps. After carefully cauterizing the tissue, the palatine tonsil was located and removed from the superior to the inferior pole. Most of the identifiable vessels supplying the tonsil were cauterized before being separated from the tonsil. Point coagulation was used to maintain hemostasis. By using point coagulation, hemostasis was maintained. To avoid bias stemming from competence, consultants performed all of these tonsillectomies.
  Arms: Bipolar electrocautery tonsillectomy group
Procedure: Cold steel dissection technique — The cold steel blunt dissection tonsillectomy was carried out under general anesthesia while the patient was in the Rose position and had an endotracheal intubation. The tonsil was retracted medially with a tonsil holding forceps, and in the upper pole, the mucosal incision was made. To protect the tonsillar pillars, a delicate dissection was performed, and the suction tip was used to stop the hemorrhage. The tonsillar fossa was packed with swabs. The other palatine tonsil was then similarly removed. Hemostasis was secured by silk ligation and bipolar electrocautery.
  Arms: Cold steel dissection group

SUMMARY:
It was intended to practically establish whether or not the relatively newer technique of tonsillectomy like bipolar electrocautery tonsillectomy has any added benefits in reducing the duration of surgery, blood loss and post-operative pain as compared with conventional cold steel dissection method. This study was done to compare the outcomes of bipolar electrocautery tonsillectomy versus cold steel dissection pediatric tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 5-13 years of age
* Both genders
* With a history of recurrent episodes of tonsillitis in the last year
* Children who had bilaterally enlarged tonsils
* No history of fever or sore throat in the last 4 weeks

Exclusion Criteria:

* Patients who had enlarged adenoids and required adenotonsillectomy
* Patients who underwent tonsillectomy after quinsy
* With a history of bleeding disorders
* Patients who showed an international normalized ratio (INR) ≥ 1.5

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Operative time | 1 hour
  Operative time was measured from the anterior pillar incision to the removal of the mouth gag.
Blood loss | up to 24 hours
  Intraoperative blood loss was measured by reading the levels given in the suction bottle at the end of surgery. The weight of dry gauze was subtracted from the wet, considering 1g=1ml.
Postoperative pain | 24 hours
  Postoperative pain was measured at regular intervals (6-hourly till 24 hours) using the Wong-Baker faces pain rating scale.12 The Wong-Baker faces pain rating scale graded pain as mild (1-3), moderate (4-6), or severe (>6).

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Ganga Ram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared with other researchers on a reasonable request.